CLINICAL TRIAL: NCT01377064
Title: Home-based Exercise for Management of HIV-associated Cardiovascular Disease
Brief Title: Home-based Exercise for Management of HIV-associated Cardiovascular Disease Risk
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00007339; 1R21NR011281 (NIH)
Record Dates: First submitted 2011-06-08; First posted 2011-06-20 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Diseases; Hyperlipidemia; Obesity
Keywords: HIV; physical activity; cardiovascular disease risk
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical activity group (Experimental): Subjects will participant in physical activity program
  Interventions: Behavioral: Physical Activity Group
- Standard care group (Active Comparator): This group will not receive a physical activity intervention
  Interventions: Other: Standard Care Group

INTERVENTIONS:
Behavioral: Physical Activity Group — 9 months of home based physical activity meeting HHS recommendations for physical activity for all americans
  Arms: Physical activity group
Other: Standard Care Group — No intervention, the group will be followed under their standard medical care.
  Arms: Standard care group

SUMMARY:
Because of advances in drug treatment, people living with HIV/AIDS (PLWHA) are living longer, but are also at greater risk for cardiovascular disease (CVD) and diabetes. Exercise and increased physical activity can reduce the risk factors for these diseases in PLWHA, but no studies have tested an at-home exercise program that would benefit low income people and others who do not have access to exercise facilities. This study will test the feasibility of an at-home exercise program for PLWHA and prepare for a full-scale intervention study, which may lead to a reduction in CVD risk among PLWHA.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Medical diagnosis of HIV-1 positive serostatus
* Sedentary lifestyle: not actively exercising ≥ 3 d•wk-1 for 20 min per session
* 18.5 kg/m2 < BMI < 40.0 kg/m2
* Stable, DHHS-approved ART regimen for previous 3 months, with HIV viral load below 75 copies/mL
* Capable of performing the required exercise regimen
* Have daily access to a telephone for approximately 10 months
* Capacity and willingness to provide informed consent and accept randomized group assignment

Exclusion Criteria:

* Individuals who have a clinical history strongly suggestive of Type 1 diabetes.
* History of serious arrythmias, cardiomyopathy, congestive heart failure, stroke or transient ischemic cerebral attacks, peripheral vascular disease with intermittent claudication, myocardial infarction, or CABG.
* Malignancies in the past 5 years, except therapeutically controlled skin cancer.
* Plans to be away > 4 weeks in the next 9 months
* Score of 5 or greater on the DAST or MAST (signifying excessive use of drugs or alcohol).
* Weight loss in excess of 10% body weight in previous 12 weeks.
* Chronic or recurrent respiratory, gastrointestinal, neuromuscular, neurological, or psychiatric conditions.
* Inflammatory-related conditions such as collagen disorders.
* Any other medical condition or disease that is life-threatening or that can interfere with or be aggravated by exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Amount of Physical Activity | 9 months
  Accelerometer data will be the primary means of determining the participants' physical activity levels. Participants will be instructed to wear the accelerometer at baseline, 4 months, and 9 months. The participants will be required to wear the accelerometer during the waking hours for seven consecutive days. Data from participants with at least four days and at least 10 hours per day will be included.

SECONDARY OUTCOMES:
Cardiorespiratory Fitness | 9 months
  Each participant will complete a graded exercise stress test (GXT) with indirect calorimetry. This test will be used to screen for abnormal physiological responses to exercise and for determining the participant's maximal ability to utilize oxygen (an index of cardiorespiratory fitness).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Citadel, Charleston, South Carolina
  - University of South Carolina, Columbia, South Carolina

REFERENCES:
- [Derived] Jaggers JR, Dudgeon W, Blair SN, Sui X, Burgess S, Wilcox S, Hand GA. A home-based exercise intervention to increase physical activity among people living with HIV: study design of a randomized clinical trial. BMC Public Health. 2013 May 24;13:502. doi: 10.1186/1471-2458-13-502. PMID 23706094